CLINICAL TRIAL: NCT05870995
Title: A Phase II Single Arm Study of Cladribine, Cytarabine, Etoposide and Venetoclax Sequential With Reduced Dose Conditioning of Fludarabine, Busulfan and Melphalan or Total Marrow Radiation for Refractory Acute Myeloid Leukemia
Brief Title: Chemotherapy CLAGE-Ven Sequential With Reduced Intensity Conditioning for Refractory Acute Myelodi Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiong HU, Head, Blood & Marrow Transplantation Center, Rui Jin Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R/R-AML-2022
Record Dates: First submitted 2023-05-13; First posted 2023-05-23 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Refractory Leukemia
Keywords: refractory AML, allogeneic stem cell transplantation
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CLAGE-VEN-RIC-Conditioning (Experimental): Cladribine: 5mg/m2 day -21 to d -17 cytarabine: 1g/m2 day -21- to d -17 etoposide: 100mg/m2 day -17 to -15 venetoclax: 100mg day-21; 200mg day -20, 400mg day -19 to day-3 Fludarabine: 30mg/m2 day -7 to -3 Busulfan: 3.2mg/kg day -6 to -5 Melphalan: 50mg/m2 day -4 to -3. or Fludarabine 30mg/m2 day -7 to -3 Total marrow irradiation day-5 to -3 PBSC: day 0
  Conditioning regimen cane delayed to in patients with ongoing active infection or work-up of donors after CLAGE-VEN chemotherapy based on clinicians' decision. Patients receiving all-HSCT in cytopenia are classified as sequential while patients with recovered CBC are considered as bridging transplantation.
  Interventions: Drug: CALGE-VEN- RIC-conditioning

INTERVENTIONS:
Drug: CALGE-VEN- RIC-conditioning — Intensive chemotherapy Cladribine-cytarabine-etoposide -venetoclax sequential with fludarabine, busulfan and melphalan or fludarabine and total marrow irradiation

SUMMARY:
The investigators developed a protocol combining chemotherapy of cladribine, cytarabine and etoposide (CLAGE) as debulking treatment sequential with reduced intensity conditioning regimen Flu-Bu to treat patients with refractory acute myeloid leukemia (AML). In this study, the aim is to further evaluate the efficacy and feasibility of the protocol with modifications: 1) reduced dose of CLAGE; 2) Reduced intensity conditioning (RIC) regimen as fludarabine, busulfan and melphalan (MBF) or total marrow irradiation (TMI); 3) Venetoclax was added to the chemotherapy and conditioning regimen.

DETAILED DESCRIPTION:
Refractory AML is associated with poor prognosis. Allogeneic stem cell transplantation is considered as the only curative therapy. Unfortunately, conventional transplantation protocol usually has high relapse rate and high nor-relapse mortality. In previous studies, the investigators established a protocol using intensive chemotherapy (cladribine, cytarabine and etoposide) to reduced the leukemia burden followed by reduced intensity conditioning regimen of Flu-Bu3 with 7 day interval. All patients received maintenance therapy. The 1-year relapse rate was less than 20% but toxicity such as lethal infection was documented in sizable part of patients. In this study, the aim is to further evaluate the efficacy and feasibility of the protocol with following modifications: 1) dose of cytarabine and etoposide are reduced to 1g/m2 and 100mg/m2 daily; 2) conditioning regimen is based on Flu-Bu2 combined with addition of melphalan (100mg/m2) or total marrow irradiation (TMI) in case of contra-indication for busulfan or melphalan; 3) Venetoclax is added to the chemotherapy and conditioning regimen. The modifications intend to reduce both the toxicities and relapse, which may turn into a benefit of disease-free survival (DFS). This is designed as a phase II multi-center prospective study to evaluate the feasibility and efficacy of the protocol.

ELIGIBILITY:
Inclusion Criteria:

* patients with refractory AML: no remission after 2 induction therapy, relapsed AML within 6 months of 1st CR, relapse AML fail to having CR after reinduction therapy, multiple relapse and refractory relapse AML
* patients with >5% bone marrow blast by morphology or by LAIP flowcytometry at enrollment
* patients with HLA-matched sibling donor, 9-10/10 matched unrelated donor or haplo-identical family donor
* patients without active infection
* informed consent provided

Exclusion Criteria:

* patients with abnormal liver function (enzyme >2N or bilirubin >2N)
* patients with abnormal renal function (Scr >1.5N)
* patients with poor cardiac function （EF<45%）

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
disease-free survival (DFS) | 2 year
  patients remain alive in remission without disease progression or relapse

SECONDARY OUTCOMES:
complete remission (CR) | day 60
  patients achieve clinical remission after transplantation
Overall survival (OS) | 2 year
  patients remain alive
non-relapse mortality (NRM) | day 100
  patients died without evidence of disease
non-relapse mortality | 2 year
  patients died without evidence of disease
relapse | 2 year
  patients fail to achieve remission or had disease relapse
GRFS | 2 year
  patients remain alive without relapse, without grade III-IV aGVHD and moderate to severe cGVHD

CONTACTS AND LOCATIONS:
Overall Officials: Chun Wang, Study Director — Shanghai Zhaxin Integrated Traditional Chinese and Western Medicine Hospital
Locations (3):
- China (3):
  - Blood & Marrow Transplantation Center, RuiJin Hospital, Shanghai, Shanghai Municipality
  - Department of Hematology, Shanghai No 6 Hospital, Shanghai
  - Shanghai ZhaXin Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No
IPD data is available only based on request to PI and study director